CLINICAL TRIAL: NCT05730426
Title: Deep Dry Needling Versus Muscle Energy Technique on Chronic Non-specific Neck Pain; a Randomized Controlled Trial.
Brief Title: Comparison Between Deep Dry Needling and Muscle Energy Technique on Chronic Non-specific Neck Pain Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haneen Mohamed Abo El-enen Ghalwash, Teaching assisstat, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003913
Record Dates: First submitted 2023-02-05; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): In addition to Transcutaneous Electrical Nerve Stimulation (TENS) (typical,100 Hz, 20 mins), Infrared (7 mins), and Exercises (Cervical Stability Exercises through activation of deep neck flexors), patients received deep dry needling on active trigger points in selected muscles (upper trapezius, levator scapulae, and sternocleidomastoid ), 3 sessions/week, for 4 weeks period.
  Interventions: Procedure: Deep dry needling
- Group B (Active Comparator): In addition to Transcutaneous Electrical Nerve Stimulation (TENS) (typical,100 Hz, 20 mins), Infrared (7 mins), and Exercises (Cervical Stability Exercises through activation of deep neck flexors), patients received muscle energy technique (post isometric relaxation) in selected muscles (upper trapezius, levator scapulae, and sternocleidomastoid ), 3 sessions/week, for 4 weeks period.
  Interventions: Procedure: Muscle energy technique
- Group C (Placebo Comparator): Patients receive Transcutaneous Electrical Nerve Stimulation (TENS) (typical,100 Hz, 20 mins), Infrared (7 mins), and Exercises (Cervical Stability Exercises through activation of deep neck flexors) , 3 sessions/week, for 4 weeks period.
  Interventions: Procedure: Neck stability exercise

INTERVENTIONS:
Procedure: Deep dry needling — Method to decrease pain and improve function in musculoskeletal disorders.
  Arms: Group A
Procedure: Muscle energy technique — Method to decrease pain and improve function in musculoskeletal disorders.
  Other Names: Post isometric relaxation
  Arms: Group B
Procedure: Neck stability exercise — Method to decrease pain and improve function in musculoskeletal disorders.
  Arms: Group C

SUMMARY:
The goal of this clinical trial is to compare between applying deep dry needling and muscle energy technique in chronic non-specific neck pain patients. Researchers will compare between deep dry needling group, muscle energy technique group and control group to see if there are change in pain, range of motion or function.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and 40 years.
2. Current neck pain.
3. Presence of at least one or two trigger points .
4. Patients are diagnosed and referred from orthopedist complaining from chronic neck pain for at least 12 weeks.
5. No clinical treatment for neck pain within the past month.
6. lacked a history of neck and shoulder myopathy, neuropathy, myelopathy and neck, torso and shoulder surgery.
7. Patients with body mass index less than 30 kg/m2.

Exclusion Criteria:

1. Patients outside the target range.
2. Neck pain associated with vertigo.
3. Osteoporosis.
4. Diagnosed psychological disorders.
5. Fibromyalgia syndrome.
6. Vertebral fractures.
7. Spinal stenosis.
8. Tumors.
9. Previous neck surgery.
10. Red flags (night pain, severe muscle spasm, loss of involuntary weight, symptom mismatch).
11. Physiotherapeutic treatment continued in the last 3 months. Any contraindications for deep dry needling such as anticoagulants, infections and bleeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity from baseline to 4 weeks after. | at baseline and after 4 weeks from the baseline.
  Visual Analogue scale (VAS)
  * A value of 0 denotes no pain, whereas a value of 1 to 3 indicates mild pain.
  * 4 to 6 denotes moderate pain.
  * 7 to 10 denotes intense pain.
Change in function from baseline to 4 weeks after. | at baseline and after 4 weeks from the baseline.
  The Neck Disability Index (NDI) The NDI questionnaire (scored out of 50) was used to measure the patient's perceived disability resulting from their neck pain. The score for each section was from 0 to 5, with 0 represented the highest level of function and 5 represented the lowest level of function. Total NDI scores were shown as a percentage. A high score corresponded to a higher degree of disability.
  * 0-4points (0-8%) no disability.
  * 5-14points (10 - 28%) mild disability.
  * 15-24points (30-48%) moderate disability.
  * 25-34points (50- 64%) severe disability.
  * 35-50points (70-100%) complete disability.
Change in cervical range of motion (ROM) in sagittal, coronal and transverse planes from baseline to 4 weeks after. | at baseline and after 4 weeks from the baseline.
  AcuAngle® Inclinometer: (Baseline® AcuAngle Inclinometer; Elmsford, NY, U.S. PAT 2194335, 2-D Functions)
Change in pain threshold from baseline to 4 weeks after. | at baseline and after 4 weeks from the baseline.
  Pain Pressure Algometer: (BASELINE 22-POUND DOLORIMETER).

CONTACTS AND LOCATIONS:
Overall Officials: Haneen M. Ghalwash, Principal Investigator — Delta University for Science and Technology
Locations (1):
- Delta University for science and technology., Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No